CLINICAL TRIAL: NCT02455635
Title: Lower Abdominal Pain During Office Hysteroscopy As A Guide In The Assessment Of Tubal Patency In Infertile Women
Brief Title: Lower Abdominal Pain During Office Hysteroscopy Can Assess Tubal Patency in Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 135
Record Dates: First submitted 2015-05-21; First posted 2015-05-28 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Infertility
Keywords: Office Hysteroscopy; tubal patency; infertility; Lower Abdominal Pain
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- women with pain (Active Comparator): women who felt pain at time of office hystroscopy at time of saline infusion and for 15 minutes after end of procedure
  Interventions: Procedure: office hystroscopy
- women without pain (Active Comparator): women who didn't feel pain at time of office hystroscopy at time of saline infusion and for 15 minutes after end of procedure
  Interventions: Procedure: office hystroscopy

INTERVENTIONS:
Procedure: office hystroscopy — Office hysteroscopythrough vaginoscopic approach was done in gynecology out-patient clinic using a 4 mm endoscopic sheath & 30 ᵒ endoscopic camera with saline distension medium using 90-100 mmHg pressure

SUMMARY:
Office hysteroscopy through vaginoscopic approach was done in gynecology out-patient clinic with saline distension medium. The presence or absence of lower abdominal pain and the side of pain were recorded. Then, transvaginal sonography within 20 minutes was done to detect the presence of free fluid in the pouch of Douglas. Then, laparoscopy with tubal chromopertubation was done.

DETAILED DESCRIPTION:
Office hysteroscopy through vaginoscopic approach was done in gynecology out-patient clinic using a 4 mm endoscopic sheath & 30 ᵒ endoscopic camera with saline distension medium using 90-100 mmHg pressure. Meanwhile, the presence or absence of lower abdominal pain and the side of pain were recorded. Then, transvaginal sonography within 20 minutes was done to detect the presence of free fluid in the pouch of Douglas.Then, laparoscopy with tubal chromopertubation was done.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women normal semen analysis

Exclusion Criteria:

* Ladies with evidence of upper or lower genital tract infections,
* presence of free fluid in the pouch of Douglas before hysteroscopy or pelvic pathology or those with cervical stenosis that required cervical dilatation prior to hysteroscopy

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
lower abdominal pain as measured by Visual Analog Scale | at time of hystroscopy till 15 minutes after end of procedure
  Pain, as measured by Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes